CLINICAL TRIAL: NCT01567098
Title: Single Incision Versus Conventional 3-Port Laparoscopic Appendectomy: A Single Center Prospective Randomized Trial
Brief Title: Single Incision Versus Conventional 3-Port Laparoscopic Appendectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Canon KO Chan, F.R.C.S. Ed., Principal Investigator, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KC/KE-12-0051
Record Dates: First submitted 2012-03-27; First posted 2012-03-30 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SILS appendectomy (Experimental): Single incision laparoscopic appendectomy
  Interventions: Procedure: single incision laparoscopic appendectomy
- 3 Ports appendectomy (Active Comparator): performing appendectomy through conventional 3 incisions on the abdomen
  Interventions: Procedure: single incision laparoscopic appendectomy

INTERVENTIONS:
Procedure: single incision laparoscopic appendectomy — performing appendectomy through a single incision in the abdomen
  Other Names: single port appendectomy; one port appendectomy; SILS

SUMMARY:
A randomized trial to study the null hypothesis:" single incision appendectomy does not take longer operation time when compared to conventional 3-port appendectomy". The study will be carried out in a tertiary referral center in Hong Kong with a catchment population of 1 million.

DETAILED DESCRIPTION:
Since the introduction of single incision laparoscopic surgery (SILS), this approach has become more popular and various case series and reports had described its feasibility in many general surgical procedures including appendectomy, cholecystectomy, and colectomy. Despite this, strong evidence in support of SILS to be equivalent or even superior to conventional multi-port approaches remain scarce, although there are case series and comparative studies with promising results in cholecystectomy and colectomy. There are many case series available stating that single incision appendectomy may be a feasible alternative to conventional approach, but may be at the expense of a longer operating time and a higher post operative wound pain score. A recent randomized trial by St. Peter et al. was the first to test the feasibility of this approach to standard 3-port approach in appendectomy in children. Under randomized settings of this trial the single incision appendectomy produced longer operating times and resulted in greater charges. However, the primary outcome measure in this trial was wound infection and the result showed no significant differences between the two approaches. The answer to whether single incision appendectomy produces a longer operating time when compared to conventional 3-port approach remained undetermined, in particular the adult population, and therefore a randomized trial design based on operating time as its primary outcome is desired.

ELIGIBILITY:
Inclusion Criteria:

* appendicitis score >5, imaging showed no complication from appendicitis

Exclusion Criteria:

* pregnancy, mentally incapacitated, previous surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
operation time | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Canon KO Chan, F.R.C.S Ed., Principal Investigator — Hospital Authority
Locations (1):
- Department of Surgery, Kowloon, Hong Kong

REFERENCES:
- [Result] Adair J, Gromski MA, Lim RB, Nagle D. Single-incision laparoscopic right colectomy: experience with 17 consecutive cases and comparison with multiport laparoscopic right colectomy. Dis Colon Rectum. 2010 Nov;53(11):1549-54. doi: 10.1007/DCR.0b013e3181e85875. PMID 20940605
- [Result] Adair J, Gromski MA, Nagle D. Single-incision laparoscopic sigmoidectomy and rectopexy case series. Am J Surg. 2011 Aug;202(2):243-5. doi: 10.1016/j.amjsurg.2010.08.034. PMID 21810504
- [Result] Agha A, Hornung M, Iesalnieks I, Glockzin G, Schlitt HJ. Single-incision retroperitoneoscopic adrenalectomy and single-incision laparoscopic adrenalectomy. J Endourol. 2010 Nov;24(11):1765-70. doi: 10.1089/end.2010.0238. Epub 2010 Sep 19. PMID 20849304
- [Result] Fujii S, Watanabe K, Ota M, Watanabe J, Ichikawa Y, Yamagishi S, Tatsumi K, Suwa H, Kunisaki C, Taguri M, Morita S, Endo I. Single-incision laparoscopic surgery using colon-lifting technique for colorectal cancer: a matched case-control comparison with standard multiport laparoscopic surgery in terms of short-term results and access instrument cost. Surg Endosc. 2012 May;26(5):1403-11. doi: 10.1007/s00464-011-2047-9. Epub 2011 Nov 20. PMID 22101420
- [Result] Raakow R, Jacob DA. Single-Incision Cholecystectomy in about 200 Patients. Minim Invasive Surg. 2011;2011:915735. doi: 10.1155/2011/915735. Epub 2011 Jul 2. PMID 22091365
- [Result] Chandler NM, Danielson PD. Single-incision laparoscopic appendectomy vs multiport laparoscopic appendectomy in children: a retrospective comparison. J Pediatr Surg. 2010 Nov;45(11):2186-90. doi: 10.1016/j.jpedsurg.2010.07.012. PMID 21034942
- [Result] Chiu CG, Nguyen NH, Bloom SW. Single-incision laparoscopic appendectomy using conventional instruments: an initial experience using a novel technique. Surg Endosc. 2011 Apr;25(4):1153-9. doi: 10.1007/s00464-010-1332-3. Epub 2010 Oct 7. PMID 20927545
- [Result] Chouillard E, Dache A, Torcivia A, Helmy N, Ruseykin I, Gumbs A. Single-incision laparoscopic appendectomy for acute appendicitis: a preliminary experience. Surg Endosc. 2010 Aug;24(8):1861-5. doi: 10.1007/s00464-009-0860-1. Epub 2010 Jan 28. PMID 20108149
- [Result] Feinberg EJ, O'Connor DJ, Feinberg ML, Vemulapalli P, Camacho D. Single-incision laparoscopic appendectomy: an early experience. Am Surg. 2011 Mar;77(3):286-9. doi: 10.1177/000313481107700315. PMID 21375838
- [Result] Goel R, Buhari SA, Foo J, Chung LK, Wen VL, Agarwal A, Lomanto D. Single-incision laparoscopic appendectomy: prospective case series at a single centre in Singapore. Surg Laparosc Endosc Percutan Tech. 2011 Oct;21(5):318-21. doi: 10.1097/SLE.0b013e3182311bd9. PMID 22002266
- [Result] St Peter SD, Adibe OO, Juang D, Sharp SW, Garey CL, Laituri CA, Murphy JP, Andrews WS, Sharp RJ, Snyder CL, Holcomb GW 3rd, Ostlie DJ. Single incision versus standard 3-port laparoscopic appendectomy: a prospective randomized trial. Ann Surg. 2011 Oct;254(4):586-90. doi: 10.1097/SLA.0b013e31823003b5. PMID 21946218
- [Result] Andersson M, Andersson RE. The appendicitis inflammatory response score: a tool for the diagnosis of acute appendicitis that outperforms the Alvarado score. World J Surg. 2008 Aug;32(8):1843-9. doi: 10.1007/s00268-008-9649-y. PMID 18553045
- [Result] Bone RC, Balk RA, Cerra FB, Dellinger RP, Fein AM, Knaus WA, Schein RM, Sibbald WJ. Definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. The ACCP/SCCM Consensus Conference Committee. American College of Chest Physicians/Society of Critical Care Medicine. Chest. 1992 Jun;101(6):1644-55. doi: 10.1378/chest.101.6.1644. PMID 1303622
- [Result] Lin YY, Shabbir A, So JB. Laparoscopic appendectomy by residents: evaluating outcomes and learning curve. Surg Endosc. 2010 Jan;24(1):125-30. doi: 10.1007/s00464-009-0691-0. PMID 19760332
- [Result] Meinke AK, Kossuth T. What is the learning curve for laparoscopic appendectomy? Surg Endosc. 1994 May;8(5):371-5; discussion 376. doi: 10.1007/BF00642433. PMID 8073350
- [Result] McKernan JB, Champion JK. Access techniques: Veress needle--initial blind trocar insertion versus open laparoscopy with the Hasson trocar. Endosc Surg Allied Technol. 1995 Feb;3(1):35-8. PMID 7757437
- [Result] Teoh AY, Chiu PW, Wong TC, Wong SK, Lai PB, Ng EK. A case-controlled comparison of single-site access versus conventional three-port laparoscopic appendectomy. Surg Endosc. 2011 May;25(5):1415-9. doi: 10.1007/s00464-010-1406-2. Epub 2010 Oct 23. PMID 20972583